CLINICAL TRIAL: NCT05748275
Title: Randomized Trial Comparing Prediction Accuracy of Two Swept Source Optical Coherence Tomography Biometers
Status: Completed | Type: Observational
Sponsor: Multack Eye Care (Other)
Responsible Party: Sponsor
Other Study IDs: 64989743
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Argos, Then IOLMaster 700: Biometry measurements first with the Argos device followed by the IOLMaster 700 device.
  Interventions: Diagnostic Test: Argos; Diagnostic Test: IOLMaster 700
- IOLMaster 700, Then Argos: Biometry measurements first with the IOLMaster 700 device followed by the Argos device.
  Interventions: Diagnostic Test: Argos; Diagnostic Test: IOLMaster 700

INTERVENTIONS:
Diagnostic Test: Argos — Biometry measurements first with the Argos device, then the IOLMaster 700 device.
Diagnostic Test: IOLMaster 700 — Biometry measurements first with the IOLMaster 700 device, then the Argos device.

SUMMARY:
To assess if the Alcon Argos Biometer utilizing the Barrett Universal II formula for IOL calculations can give a non-inferior outcome when compared to the Zeiss IOL master 700 utilizing the (PCA) with the Barrett Universal II (TK) formula, when comparing the (mean absolute prediction error of the predicted target spherical equivalencies).

ELIGIBILITY:
Inclusion Criteria:

* Age: 50-85 years old
* Clinically Significant Cataracts that interfere with daily activities
* Patient is able to understand and able to consent to informed consent
* Patient is able to come to all postoperative visits and agrees to follow up at 30 days -2/+14 days
* Patient undergoing cataract surgery, with implantation of the Alcon SN60WF lens in the capsular bag.

Exclusion Criteria:

* Axial Length < 22.00 and > 26.00
* Corneal Astigmatism > +1.00 Diopters
* CCTS: < 490 and > 600
* Prior Refractive Surgery: RK, PRK, LASIK, INTACTS
* History of contact lens use: Soft lenses within 2 months of surgery, RGP within 60 months of surgery
* Corneal Disease: Keratoconus, Corneal Dystrophies, Any prior corneal Surgery, Prior infections
* Retinal Disease: Macular Pathology, CSCR, CME, Macular Degeneration, Drusen, Retinal Detachment, TPPV, SB, prior IVT, Prior PRP or Focal Laser, Diabetic Retinopathy
* History of Uveitis
* POAG: Undergoing any concomitant MIGS procedure- iStent, Omni, iTrack, Hydrus, etc
* Enrollment in any prior clinical trial within 2 years
* Systemic Disease that in the investigator's opinion may affect outcome
* Currently Pregnant or Breastfeeding
* Severe Dry Eye
* Tear Osmolarity > 320mOsms/L (Moderate)
* Any Surgical Complication(s)
* IOL implanted outside of the capsular bag /capsular damage /weakness /CTR placement

Ages: 50 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults presenting with clinically significant cataracts.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Multack, D.O., Principal Investigator — Multack Eye Care
Locations (1):
- Multack Eye Care, Frankfort, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Argos, Then IOLMaster 700 | IOLMaster 700, Then Argos
Started | 40; 40 Eyes | 40; 40 Eyes
Completed | 40; 40 Eyes | 40; 40 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean Absolute Prediction Error (D)
Time Frame: 1 month postoperatively
Measure: Mean (Standard Deviation); unit: diopters
Groups:
- Argos: Biometry measurements with the Argos device.
- IOLMaster 700: Biometry measurements with the IOLMaster 700 device.
Arm/Group | Argos | IOLMaster 700
Number analyzed (Participants) | 80 | 80
diopters | 0.21 (0.25) | 0.25 (0.24)

2. Secondary Outcome: Percentage of Eyes With Absolute Prediction Error 0.5 D or Less
Time Frame: 1 month postoperatively
Measure: Number; unit: percent
Units Other Than Participants: Eyes
Groups:
- Argos: Biometry measurements first with the Argos device.
- IOLMaster 700: Biometry measurements first with the IOLMaster 700 device.
Arm/Group | Argos | IOLMaster 700
Number analyzed (Participants) | 80 | 80
Number analyzed (Eyes) | 80 | 80
percent | 91 | 88

3. Secondary Outcome: Median Absolute Prediction Error (D)
Time Frame: 1 month postoperatively
Measure: Median (Inter-Quartile Range); unit: diopters
Arm/Group | Argos | IOLMaster 700
Number analyzed (Participants) | 80 | 80
diopters | 0.14 [0.06 to 0.25] | 0.19 [0.09 to 0.29]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Argos | IOLMaster 700
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT05748275/Prot_SAP_000.pdf